CLINICAL TRIAL: NCT05837910
Title: Radicle™ Calm 2: A Randomized, Double-Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Feelings of Anxiety, Stress, and Other Health Outcomes
Brief Title: Radicle Calm 2: A Study of Health and Wellness Products on Feelings of Anxiety, Stress, and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2302
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' study product assignment. Participants are blinded to the study product they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Placebo Control 1 (Placebo Comparator): Calm Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Active Product 1.1 (Experimental): Calm Product Form 1 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 1.1 Usage
- Active Product 1.2 (Experimental): Calm Product Form 1 - active product 2
  Interventions: Dietary Supplement: Calm Active Study Product 1.2 Usage
- Active Product 1.3 (Experimental): Calm Product Form 1 - active product 3
  Interventions: Dietary Supplement: Calm Active Study Product 1.3 Usage
- Placebo Control 2 (Placebo Comparator): Calm Product Form 2 - control
  Interventions: Dietary Supplement: Placebo Control Form 2
- Active Product 2.1 (Experimental): Calm Product Form 2 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 2.1 Usage
- Placebo Control 3 (Placebo Comparator): Calm Product Form 3 - control
  Interventions: Dietary Supplement: Placebo Control Form 3
- Active Product 3.1 (Experimental): Calm Product Form 3 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 3.1 Usage
- Placebo Control 4 (Placebo Comparator): Calm Product Form 4 - control
  Interventions: Dietary Supplement: Placebo Control Form 4
- Active Product 4.1 (Experimental): Calm Product Form 4 - active product 1
  Interventions: Dietary Supplement: Calm Active Study Product 4.1 Usage

INTERVENTIONS:
Dietary Supplement: Calm Active Study Product 1.1 Usage — Participants will use their Radicle Calm Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Calm Active Study Product 1.2 Usage — Participants will use their Radicle Calm Active Study Product 1.2 as directed for a period of 6 weeks.
  Arms: Active Product 1.2
Dietary Supplement: Calm Active Study Product 1.3 Usage — Participants will use their Radicle Calm Active Study Product 1.3 as directed for a period of 6 weeks.
  Arms: Active Product 1.3
Dietary Supplement: Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Placebo Control Form 2 — Participants will use their Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Calm Active Study Product 2.1 Usage — Participants will use their Radicle Calm Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Placebo Control Form 3 — Participants will use their Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Calm Active Study Product 3.1 Usage — Participants will use their Radicle Calm Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Placebo Control Form 4 — Participants will use their Placebo Control Form 4 as directed for a period of 6 weeks.
  Arms: Placebo Control 4
Dietary Supplement: Calm Active Study Product 4.1 Usage — Participants will use their Radicle Calm Active Study Product 4.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1

SUMMARY:
A randomized, double-blinded, placebo-controlled study assessing the impact of health and wellness products on feeling of anxiety, stress, and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for less anxiety or stress, (2) indicate an interest in taking a health and wellness product to potentially help their feelings of anxiety or stress, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses fewer feelings of anxiety or stress as a primary desire
* Selects feelings of anxiety or stress, looking to improve their feelings of anxiety or stress, and/or reduce reliance on medications as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address
* The calculated validated health survey (PRO) measurement result is less than mild severity/impairment
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in a clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy, immunotherapy, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied: anticoagulants, a medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, or MAOIs (monoamine oxidase inhibitors)
* Reports a diagnosis of heart disease when a known contraindication exists for any of the active ingredients studied: NYHA (New York Heart Association) Class III or IV congestive heart failure, Atrial fibrillation, Uncontrolled arrhythmias

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3853 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Change in feelings of anxiety | 6 weeks
  Mean difference in feelings of anxiety score as assessed by Patient Reported Outcome Measurement System (PROMIS) Anxiety 8A (scale 8-40; where lower scores correspond to less feelings of anxiety)

SECONDARY OUTCOMES:
Change in stress | 6 weeks
  Mean difference in stress score as assessed by National Institutes of Health (NIH) Toolbox Perceived Stress Survey (scale 10-50; where lower scores correspond to less stress)
Change in cognitive function | 6 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognition Function 4A (scale 4-20; where lower scores correspond to poorer cognitive function)
Change in sleep | 6 weeks
  Mean difference in sleep score as assessed by PROMIS Sleep Disturbance 4A (scale 4-20; where lower scores correspond to better sleep quality/less sleep disturbance)
Change in mood (emotional distress) | 6 weeks
  Mean difference in mood score as assessed by PROMIS Emotional Distress-Depression 4A (scale 4-20; where lower scores correspond to lower levels of emotional distress)
Change in libido | 6 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; where lower scores correspond to less interest in sexual activity)
Minimal clinically important difference (MCID) in feelings of anxiety | 6 weeks
  Likelihood of achieving a MCID in sleep disturbance, as measured by PROMIS Anxiety 8A (scale 8-40; where lower scores correspond to less feelings of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com